CLINICAL TRIAL: NCT03142685
Title: Pilot Randomized Control Trial of Necrotizing Enterocolitis Screening Using Abdominal Radiograph Versus Bowel Ultrasound Plus Abdominal Radiograph in Congenital Heart Disease Patients
Brief Title: Utility of Bowel Ultrasound in Diagnosing Necrotizing Eneterocolitis in Congenital Heart Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Sherwin Chan, Pediatric Radiologist, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16010050
Record Dates: First submitted 2017-04-26; First posted 2017-05-05 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Enterocolitis, Necrotizing; Congenital Heart Disease
Keywords: NEC; Bowel Ultrasound; CHD
MeSH Terms: conditions — Enterocolitis, Necrotizing; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: This is a prospective pilot randomized control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm B: Kub + Bowel US (Experimental): Subjects clinical suspected of NEC whom are randomized into Arm B at time of consent will receive a bowel ultrasound q24 for 48 hours and a KUB q12 for 48 hours.
  Interventions: Device: Bowel Ultrasound
- Arm A: KUB Only (No Intervention): Subjects clinical suspected of NEC whom are randomized into Arm A at time of consent will receive a KUB q12 for 48 hours. This is the current standard-of-care procedures.

INTERVENTIONS:
Device: Bowel Ultrasound — Subjects randomized to Arm B will undergo a bowel ultrasound q24 for 48 hours after time of clinical suspicion of NEC. This is in addition to the standard of care KUBs which patients in both arms will get.
  Arms: Arm B: Kub + Bowel US

SUMMARY:
To evaluate the feasibility of performing a randomized pilot control trial of two diagnostic screening strategies for necrotizing enterocolitis in patients with congenital heart disease. Measures to evaluate will be the ability to obtain consent from patients, percentage of eligible patients that are able to be recruited, coordination of providers, estimation of degree of crossover and ability to perform the screening exams per protocol.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is the most common bowel disease in premature and low birth weight neonates. NEC is defined by the loss of mucosal integrity of the bowel wall enabling bacteria and other toxins to permeate into the bowel causing ischemia and necrosis which can lead to bowel perforation and sepsis. NEC can result in substantial morbidity and mortality and prolonged hospital and ICU stays.

Studies have shown that full-term neonates with congenital heart disease (CHD) are 3.7 to 6.3 times as likely to develop NEC compared with other premature neonates. The overall incidence of CHD is up to 12-14 per 1,000 live births and the incidence of NEC in patients with severe CHD is up to 10%. Patients with CHD have diastolic hypoperfusion causing inadequate blood circulation which can increase their risk of developing NEC. Treatment of NEC is often dependent on the clinical severity of the patient. Conservative treatment can be done in early stages of suspicion of NEC, while more severe NEC requires resection of the necrotic bowel. The current standard of care for diagnosis of NEC is based upon clinical suspicion, laboratory values and imaging characteristics found on an abdominal radiograph. Clinicians use the Modified Bells Staging Criteria (Appendix A) to diagnose patients with suspected NEC. Clinical manifestations often include abdominal bloating, feeding intolerance, constipation, emesis, ileus, and/or occult or frank blood in stool.

In the past, abdominal radiography has been scored on a standard scale that correlated with outcomes. Duke University Medical Center developed a standardized ten-point radiographic scale, the Duke Abdominal Assessment Scale (DAAS) and was proven to be directly proportional to the severity of NEC on patients that underwent surgery. Abdominal radiographs are assessed for gas pattern, bowel distention, location and features, pneumatosis (gas in bowel wall), portal venous gas and pneumoperitoneum (free air in peritoneal cavity) to indicate the level of suspicion of NEC . The use of abdominal radiographs is the most common assessment for suspected NEC in infants, however, there have been recent studies done on the utility of bowel ultrasound to aid in early diagnosis of NEC due to the ability to evaluate peristalsis, echogenicity and thickness of bowel wall, pneumatosis and the capability of doing color Doppler to evaluate blood perfusion. A University of Toronto study used ultrasound to assess bowel perfusion with color Doppler in neonates and found a correlation between absence of bowel wall perfusion and the increased severity of NEC on surgical pathology . Although there are similar signs found between abdominal radiography and bowel ultrasound, some of the more severe features such as, pneumoperitoneum, were found to be more sensitive on bowel ultrasound, thus potentially leading to more definitive treatment . Currently, there is no good study evaluating whether the use of bowel ultrasound affects clinical outcomes in patients with CHD over the use of abdominal radiography alone.

The use bowel ultrasound has yet to be adopted in the setting of suspicion for NEC at our institution. This is primarily due to the lack of expertise of the ultrasound technologists, radiologists and clinicians. With literature dating back to 2005 supporting the use of bowel ultrasound in diagnosis of severity of NEC, a high volume of CHD patients at our institution as well as new radiologists trained in bowel ultrasound, we would like to see if a regimen involving combined ultrasound and radiograph screening for NEC would make a difference in clinical outcomes (morbidity, mortality, and length of stay (LOS)) compared with radiograph screening alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 0-6 months with CHD
* Completed one or more cardiac surgeries for CHD
* Clinicians are suspicious for NEC and order an abdominal radiograph for screening.

Exclusion Criteria:

* Patients with isolated PDA or PFO congenital cardiac abnormalities
* Unable to ultrasound the bowel (eg. gut in silo)
* Prior heart transplant

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Days NPO due to NEC concern | From the date of enrollment to the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 500 days.
  The number of days that a patient has no enteral feedings due to concern for necrotizing enterocolitis.

SECONDARY OUTCOMES:
ICU length of stay | From the date of enrollment to the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 500 days.
  Days in the ICU during the current hospitalization
Hospital length of stay | From the date of enrollment to the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 500 days.
  Days in the hospital during the current hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin S Chan, MD PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] M. Epelman, A. Daneman, D. Podeberesky, L. Averill, K. Darge, paper presented at the Radiological Society of North America, Chicago, 2015.
- [Result] Epelman M, Daneman A, Navarro OM, Morag I, Moore AM, Kim JH, Faingold R, Taylor G, Gerstle JT. Necrotizing enterocolitis: review of state-of-the-art imaging findings with pathologic correlation. Radiographics. 2007 Mar-Apr;27(2):285-305. doi: 10.1148/rg.272055098. PMID 17374854
- [Result] Staryszak J, Stopa J, Kucharska-Miasik I, Osuchowska M, Guz W, Blaz W. Usefulness of ultrasound examinations in the diagnostics of necrotizing enterocolitis. Pol J Radiol. 2015 Jan 1;80:1-9. doi: 10.12659/PJR.890539. eCollection 2015. PMID 25574248
- [Result] Pickard SS, Feinstein JA, Popat RA, Huang L, Dutta S. Short- and long-term outcomes of necrotizing enterocolitis in infants with congenital heart disease. Pediatrics. 2009 May;123(5):e901-6. doi: 10.1542/peds.2008-3216. PMID 19403484
- [Result] McElhinney DB, Hedrick HL, Bush DM, Pereira GR, Stafford PW, Gaynor JW, Spray TL, Wernovsky G. Necrotizing enterocolitis in neonates with congenital heart disease: risk factors and outcomes. Pediatrics. 2000 Nov;106(5):1080-7. doi: 10.1542/peds.106.5.1080. PMID 11061778
- [Result] Motta C, Scott W, Mahony L, Koch J, Wyckoff M, Reisch J, Burchfield PJ, Brion LP. The association of congenital heart disease with necrotizing enterocolitis in preterm infants: a birth cohort study. J Perinatol. 2015 Nov;35(11):949-53. doi: 10.1038/jp.2015.96. Epub 2015 Aug 6. PMID 26248130
- [Result] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Result] Becker KC, Hornik CP, Cotten CM, Clark RH, Hill KD, Smith PB, Lenfestey RW. Necrotizing enterocolitis in infants with ductal-dependent congenital heart disease. Am J Perinatol. 2015 Jun;32(7):633-8. doi: 10.1055/s-0034-1390349. Epub 2014 Dec 8. PMID 25486286
- [Result] Walsh MC, Kliegman RM. Necrotizing enterocolitis: treatment based on staging criteria. Pediatr Clin North Am. 1986 Feb;33(1):179-201. doi: 10.1016/s0031-3955(16)34975-6. PMID 3081865
- [Result] Kim WY, Kim WS, Kim IO, Kwon TH, Chang W, Lee EK. Sonographic evaluation of neonates with early-stage necrotizing enterocolitis. Pediatr Radiol. 2005 Nov;35(11):1056-61. doi: 10.1007/s00247-005-1533-4. Epub 2005 Aug 3. PMID 16078076
- [Result] Coursey CA, Hollingsworth CL, Gaca AM, Maxfield C, Delong D, Bisset G 3rd. Radiologists' agreement when using a 10-point scale to report abdominal radiographic findings of necrotizing enterocolitis in neonates and infants. AJR Am J Roentgenol. 2008 Jul;191(1):190-7. doi: 10.2214/ajr.07.3558. PMID 18562745
- [Result] Faingold R, Daneman A, Tomlinson G, Babyn PS, Manson DE, Mohanta A, Moore AM, Hellmann J, Smith C, Gerstle T, Kim JH. Necrotizing enterocolitis: assessment of bowel viability with color doppler US. Radiology. 2005 May;235(2):587-94. doi: 10.1148/radiol.2352031718. PMID 15858098